CLINICAL TRIAL: NCT05885321
Title: Exploring the Correlation Between Post Traumatic Stress Disorder, Perceived Stress and Scar Pruritus in Burn Patients
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202212108RINC
Record Dates: First submitted 2023-02-21; First posted 2023-06-01 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2023-12

CONDITIONS: Burns; Scar Pruritus; Post Traumatic Stress Disorder; Perceived Stress
MeSH Terms: conditions — Burns; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Pruritus, post traumatic stress disorder and perceived stress are common issues in burn patients. The correlation between the three is unclear so far.

This study will collect data among adult patients with hypertrophic scars 21 days after the burn event has occurred. Using a Chinese version of the 5D itch scale,Chinese version of the posttraumatic diagnostic scale and Perceived Stress Scale to investigate self-reported postburn pruritus,post traumatic stress disorder and perceived stress. The patients will be wearing the smart watch for one month to collect data on their stress levels. This data will be used to analyze the correlation between posttraumatic stress syndrome, perceived stress and scar pruritus. There will be two rounds of data collection. The first will be when the smart watch is issued to patients, and the second will be at the end of the one month period.

ELIGIBILITY:
Inclusion Criteria:

* Patients with hypertrophic scars 21 days after the burn event occurred
* Adult patients over 18 years old
* Patients without serious mental disorders, and are able to express themselves in Chinese with clear consciousness.
* The patient has no open wound on the wrist and is able to wear the smart watch continuously for one month

Exclusion Criteria:

* Patients with first-degree burns
* Non-traumatic electrical burns

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Patients with hypertrophic scars 3 months after the burn event occurred
  * Adult patients over 18 years old
  * Patients without serious mental disorders, and are able to express themselves in Chinese with clear consciousness.
  * The patient has no open wound on the wrist and is able to wear the smart watch continuously for one month
Sampling Method: Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2023-03-06 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
the Chinese version of the 5D itch scale | up to one months
  mmeasure the scar pruritus in burn patients,This scale including 5 domains: duration, degree, direction, disability and distribution. The duration, degree and direction domains each included one item, while the disability domain had four items. All items of the first four domains were measured on a five-point Likert scale.The distribution domain included 16 potential locations of itch,The scores of each of the five domains are achieved separately and then summed together to obtain a total 5-D score. 5-D scores can potentially range between 5 (no pruritus) and 25 (most severe pruritus).
Chinese version of Perceived Stress Scale | up to one months
  measure the Perceived Stress in burn patients,The Perceived Stress Scale consists of 14 items ,The scale can cluster into two subscales: negative subscale (items 1,2,3,8,11,12 and 14) and positive subscale (items 4,5,6,7,9,10 and 13), Each item is rated on a five-point scale from 0 = 'never' to 4 = 'very often', covering the preceding month
Chinese version of the post traumatic diagnostic scale for DSM-5 | up to one months
  measure the post traumatic stress in burn patients,a cutoff score of 28 for identifying a probable PTSD diagnosis
garmin_Vivosmart 3 | up to one months
  measure the Stress in burn patients By analyzing heart rate variability, a device can provide an assessment of an individual's overall general life stress. The stress level is measured on a scale from 0 to 100, where 0 to 25 represents a resting state, 26 to 50 indicates low stress, 51 to 75 signifies medium stress, and 76 to 100 indicates a high stress state. This device enables users to view their all-day stress levels as well as observe long-term trends.

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No